CLINICAL TRIAL: NCT01152606
Title: An Observational Study of Cardiac Events in Patients With HER2 Positive Early Breast Cancer Treated With Herceptin
Brief Title: A Study of Cardiac Safety in Patients With HER2 Positive Early Breast Cancer Treated With Herceptin
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: BO20652
Record Dates: First submitted 2010-06-28; First posted 2010-06-29 (Estimated); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort
  Interventions: Drug: trastuzumab [Herceptin]

INTERVENTIONS:
Drug: trastuzumab [Herceptin] — There is no planned investigational product or a treatment regimen prescribed by this protocol. Decision about a treatment regimen will be made according to the local practice and in the best interest of individual patients.

SUMMARY:
This is a single cohort observational safety study. All patients will be treated and monitored according to the local clinical practice. No additional procedures/patient visits in comparison with the usual clinical practice are planned for the study. Data will be collected from centre's medical records for up to 5 years or death.

ELIGIBILITY:
Inclusion Criteria:

* All patients who are considered candidates to receive Herceptin for this indication

Exclusion Criteria:

* Patients for whom Herceptin is contraindicated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HER2-positive Breast Cancer
Sampling Method: Probability Sample
Enrollment: 3942 (Actual)
Dates: Start 2007-08-30 (Actual); Primary Completion 2016-05-31 (Actual); Study Completion 2016-05-31 (Actual)

PRIMARY OUTCOMES:
Incidence of symptomatic congestive heart failure\n(CHF) using New York Heart Association class II, III and IV, and cardiac death | On treatment and up to 5 years follow-up

SECONDARY OUTCOMES:
Time to onset and the time to recovery of symptomatic congestive heart failure | On treatment and up to 5 years follow-up
Incidence of asymptomatic cardiac failure and other significant cardiac conditions | On treatment and up to 5 years follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (205):
- Austria (15):
  - Lkh-Univ. Klinikum Graz; Klinik Für Gynäkologie, Graz
  - LKH-UNIV. KLINIKUM GRAZ; Klinische Abteilung für Onkologie, Graz
  - Lhk Klagenfurt; Abt. Für Gynäkologie, Klagenfurt
  - LKH Hochsteiermark; Abt. für Innere Medizin, Leoben
  - Ordensklinikum Linz Barmherzige Schwestern; Abt. fur Innere Medizin 1, Linz
  - Lhk Feldkirch; Interne Medizin Abt., Rankweil
  - Lkh Salzburg - Univ. Klinikum Salzburg; Iii. Medizinische Abt., Salzburg
  - A. Ö. Krankenhaus Der Barmherzigen Brüder; Abt. Für Chirurgie, Sankt Veit an der Glan
  - A.Ö. Lhk; Ii. Medizinische Abt. Mit Schwerpunkt Gaströnter. & Onkologie, Steyr
  - Krankenanstalt Rudolfstiftung; I. Med. Abt., Vienna
  - Medizinische Universität Wien; Univ.Klinik für Frauenheilkunde - Klinik für Gynäkologie, Vienna
  - Medizinische Universität Wien; Univ.Klinik für Innere Medizin I, Vienna
  - Wilhelminenspital; I. Medizinische Abt., Vienna
  - Lhk Vöcklabruck; Ii. Interne Abt., Vöcklabruck
  - Klinikum Kreuzschwestern Wels; Iv. Interne Abt., Wels
- Belgium (16):
  - ZNA Middelheim, Antwerp
  - CH EpiCURA Site Louis Caty, Baudour
  - AZ KLINA, Brasschaat
  - AZ Sint Jan, Bruges
  - HIS (Etterbeek Ixelles), Brussels
  - Hospital Erasme; Neurologie, Brussels
  - Cliniques Universitaires St-Luc, Brussels
  - UZ Antwerpen, Edegem
  - AZ Groeninge (Kennedylaan), Kortrijk
  - CHU Sart-Tilman, Liège
  - Clinique Ste-Elisabeth, Namur
  - Clinique St Pierre asbl, Ottignies
  - AZ Delta (Campus Wilgenstraat), Roeselare
  - AZ Nikolaas (Sint Niklaas), Sint-Niklaas
  - AZ Turnhout Sint Elisabeth, Turnhout
  - Sint Augustinus Wilrijk, Wilrijk
- Germany (69):
  - Studienzentrum Aschaffenburg, Aschaffenburg
  - Internist; Praxis Für Haemotologie & Onkologie, Bad Soden
  - Brustzentrum Bassum, Bassum
  - Onkologische Schwerpunktpraxis Kurfürstendamm, Berlin
  - Praxis Dr. Schoenegg, Berlin
  - DRK Kliniken Berlin Köpenick, Frauenklinik, Berlin
  - Praxis Dr Geuther, Berlin
  - Onkologische Schwerpunktpraxis Bielefeld; Haemotologie & Internistische onkologie, Bielefeld
  - Medizinisches Versorgungszentrum Bonn, Bonn
  - Universitätsklinikum Bonn; Zentrum für Geburtshilfe und Frauenheilkunde, Bonn
  - Gemeinschaftspraxis Für Haematologie/Onkologie, Cologne
  - Uniklinik Köln; Klinik Für Frauenheilkunde, Cologne
  - Med. Versorgungszentrum Filiale Donauwörth Onkologisches Zentrum, Donauwörth
  - Onkologisches Zentrum; Oncology, Donauwörth
  - St. Johannes Hospital, Dortmund
  - Praxis im Elbcenter 1 in Dresden-Pieschen; Dr. med. Thomas Goehler & Dipl.-Med. Steffen Doerfel, Dresden
  - BAG Freiberg-Richter, Jacobasch, Illmer, Wolf, Dresden
  - Universitätsklinikum "Carl Gustav Carus"; Frauenheilkunde und Geburtshilfe, Dresden
  - Universitätsklinikum Düsseldorf; Frauenklinik, Düsseldorf
  - Kreisklinik Ebersberg; Abteilung für Gynäkologie & Geburtshilfe, Ebersberg
  - Universitätsklinikum Erlangen; Frauenklinik, Erlangen
  - St Antonius Hospital; Frauenklinik, Eschweiler
  - Uniklinik Essen; Gynäkologie, Essen
  - Hämatologisch-Onkologische Gemeinschaftspraxis am Bethanien-Krankenhaus, Frankfurt am Main
  - Praxis für Interdisziplinäre Onkologie und Hämatologie GbR, Freiburg im Breisgau
  - Klinikum Fulda gAG; Frauenklinik, Fulda
  - Klinikum St. Georg GmbH; Franziskus-Hospital Harderberg; Klinik für Gynaekologie und Geburtshilfe, Georgsmarienhütte
  - Wilhelm-Anton-Hospital Klinik f.Hämatologie und internistische Onkologie, Goch
  - Martin-Luther-Universität Halle-Wittenberg, Halle
  - Universitätsklinikum Hamburg-Eppendorf; Frauenklinik, Hamburg
  - Kooperatives Mammazentrum Hamburg Krankenhaus Jerusalem, Hamburg
  - Praxis Harburger Ring, Hamburg
  - Iorc-Innovation Onkologie& Research& Consulting Gmbh; Praxis Lerchenfeld Hamburg, Hamburg
  - Dres. Sigrun Müller-Hagen Mathias Bertram und Ulrich Stein, Hamburg
  - SANA Klinikum Hameln-Pyrmont; Frauenklinik / Brustzentrum, Hamelin
  - Diakovere Henriettenstift, Frauenklinik, Hanover
  - Medizinische Hochschule Zentrum Frauenheilkunde Abt.Gynäkologische Onkologie, Hanover
  - Stiftung Kathol. Krankenhaus Marienhospital Herne Klinik Mitte Frauenklinik, Herne
  - Universitaetsklinikum des Saarlandes; Klinik f. Frauenheilkunden und Geburtshilfe, Homburg/Saar
  - Universitätsklinikum Jena; Klinik und Poliklinik für Frauenheilkunde und Fortpflanzungsmedizin, Jena
  - Westpfalz-Klinikum GmbH; Klinik für Frauenheilkunde und Geburtshilfe, Kaiserslautern
  - Gemeinschaftspraxis Dr. Siehl & Dr. Soeling, Kassel
  - Systemedic Frauenarzte Pruener Gang, Kiel
  - Asklepios Klinik; Abt. Gynäkologie, Langen
  - Klinik Lippe Lemgo; Medizinische Klinik II/Haematoonkologie, Lemgo
  - Universitätsklinikum Schleswig-Holstein / Campus Lübeck; Klinik für Frauenheilkunde und Geburtshilfe, Lübeck
  - Onkologische Gemeinschaftspraxis, Magdeburg
  - Universitätsmedizin Mainz; Klinik u. Poliklinik f. Geburtshilfe u. Frauenheilkunde, Mainz
  - Universitätsklinikum Marburg; Gynäkologie, Marburg
  - Ev. Krankenhaus, Mülheim
  - Gemeinschaftspraxis für Hämatologie und Onkologie, Münster
  - Praxis Für Haematologie & Onkologie Dr. B. Otremba, Oldenburg
  - Praxis Frau Dr. Schwarz, Oranienburg
  - Klinikum Passau; 2. Medizinische Klinik; Onkologie und Hämatologie, Passau
  - Krankenhaus Rheinfelden; Frauenklinik, Rheinfelden
  - Agaplesion Diakonieklinikum Rotenburg, Rotenburg (Wümme)
  - Caritas Klinik St. Theresia -Frauenklinik Brustzentrum, Saarbrücken
  - Praxis Dr. Wagner, Saarbrücken
  - Klinik Saarbrücken Ggmbh; Brustzentrum, Saarbrücken
  - DRK Krankenhaus Saarlouis; Kooperatives Brustzentrum, Saarlouis
  - Marienkrankenhaus Abt. Gynäkologie und Geburtshilfe, Saint Wendel
  - MVZ für Hämatologie, Onkologie, Strahlentherapie und Palliativmedizin -; Klinik Dr. Hancken, Stade
  - Johanniter-Krankenhaus, Stendal
  - Klinik Der Hansestadt Stralsund Gmbh; Frauenklinik, Stralsund
  - Klinikum Traunstein, Traunstein
  - Klinikum Mutterhaus der Borromaeerinnen gGmbH; Haematologie/Onkologie, Trier
  - Katharinen-Hospital gGmbH, Unna
  - Kliniken Nordoberpfalz; Klinikum Weiden; Brustzentrum, Weiden
  - Gemeinschaftspraxis Hämatologie / Onkologie, Wiesbaden
- Hungary (4):
  - Semmelweis Egyetem Onkologiai Központ, Budapest
  - Municipal Hospital of Uzsoki Utca; Centre of Oncoradiology, Budapest
  - Josa Andras Korhaz; Dept of Oncoradiology, Nyíregyháza
  - Vas Megyei Markusovszky Korhaz ; Pulmonology, Szombathely
- Italy (58):
  - Policlinico Ospedaliero Ss Annunziata; U.O. Di Clinica Oncologica, Chieti, Abruzzo
  - Ospedale Vito Fazzi; Div. Oncoematologia, Lecce, Apulia
  - IRCCS Ospedale Casa Sollievo Della Sofferenza; Oncologia, San Giovanni Rotondo, Apulia
  - Ospedale San Carlo; Day Hospital Oncologia Medica, Potenza, Basilicate
  - Ospedale Oncologico Regionale; U.O. Oncologia Medica Ed Ematologia, Rionero in Vulture, Basilicate
  - Az. Osp. Pugliese; Dh Oncologico, Catanzaro, Calabria
  - Az. Osp. Mariano Santo; Centro Oncologico, Cosenza, Calabria
  - Azienda Ospedaliera S.G. Moscati; Division of Medical Oncology, Avellino, Campania
  - Az. Osp. Cardarelli; Divisione Di Oncologia, Napoli, Campania
  - Ist. Uni Federico Ii; Divisione Di Oncologia Medica - Dpt. Di Medicina Interna, Napoli, Campania
  - Istituto Tumori Fondazione Pascale; Endocrinologia Oncologica, Napoli, Campania
  - Ospedale S. Gennaro; Oncologia Medica, Napoli, Campania
  - Az. Osp. S. Orsola Malpighi; Istituto Di Oncologia Seragnoli, Bologna, Emilia-Romagna
  - Opspedale Morgagni - Pierantoni; Dept. Di Oncologia Medica, Meldola, Emilia-Romagna
  - Ospedale Provinciale Santa Maria delle Croci, Ravenna, Emilia-Romagna
  - Irccs Centro Di Riferimento Oncologico (CRO); Dipartimento Di Oncologia Medica, Aviano, Friuli Venezia Giulia
  - Centro Soc. Oncologico, Azienda Sanitaria Universitaria Integrata Trieste; CENTRO ONCOLOGICO, Trieste, Friuli Venezia Giulia
  - Ospedale S. Maria Goretti; Divisione Di Oncologia Medica, Latina, Lazio
  - Ospedale San Giacomo in Augusta; Reparto Oncologia, Rome, Lazio
  - Policlinico Universitario Campus Biomedico; Uoc Oncologia Medica, Rome, Lazio
  - Azienda Complesso Ospedaliero S. Filippo Neri; Divisione Di Oncologia Medica, Rome, Lazio
  - Istituto Regina Elena; Oncologia Medica A, Rome, Lazio
  - Policlinico Militare Di Roma; Reparto Di Oncologia, Rome, Lazio
  - IRCCS Istituto Nazionale Per La Ricerca Sul Cancro (IST); Oncologia Medica A, Genoa, Liguria
  - Ospedale S. Andrea Est Felettino; Oncologia Medica, La Spezia, Liguria
  - Asst Papa Giovanni XXIII; Oncologia Medica, Bergamo, Lombardy
  - Az. Osp. Spedali Civili; Divisione Di Oncologia - Iii Medicina, Brescia, Lombardy
  - Ospedale Di Casalpusterlengo; Day Hospital Oncologico, Casalpusterlengo, Lombardy
  - Ospedale Valduce; Dept. Di Oncologia Medica, Como, Lombardy
  - ASST DI LECCO; Oncologia Medica, Lecco, Lombardy
  - ASST OVEST MILANESE; Oncologia Medica, Legnano, Lombardy
  - Az. Osp. Carlo Poma; Divisione Di Oncologia Medica, Mantova, Lombardy
  - Istituto Europeo Di Oncologia, Milan, Lombardy
  - Asst Santi Paolo E Carlo; Unita Operativa Di Oncologia Medica, Milan, Lombardy
  - Fondazione Salvatore Maugeri; Divisione Di Oncologia Medica, Pavia, Lombardy
  - Fondazione Salvatore Maugeri; Servizio Di Prevenzione Oncologica, Pavia, Lombardy
  - Irccs Policlinico S. Matteo - Uni Pavia; Clinica Medica I Div. Med. Int. Onc. Medica E Gastroent., Pavia, Lombardy
  - Ospedale Di Circolo; Centro Di Senologia, Varese, Lombardy
  - Fondazione Del Piemonte Per L'oncologia Ircc Di Candiolo; Dipartimento Oncologico, Candiolo, Piedmont
  - Ospedale Degli Infermi Di Biella; Reparto Oncologia Medica, Ponderano (BI), Piedmont
  - A.O. Città della Salute e della Scienza - Presidio Molinette; divisione oncologia medica, Turin, Piedmont
  - Ospedale Sant'Anna - Uni Di Torino; Unita Di Oncologia Ginecologica, Turin, Piedmont
  - A.O.U. Cagliari-P.O. Monserrato;U.O. Oncologia, Cagliari, Sardinia
  - Azienda Ospedaliero Universitaria Di Sassari;Oncologia, Sassari, Sardinia
  - Centro Catanese Di Oncologia; Oncologia Medica, Catania, Sicily
  - Az. Osp. M. Ascoli G. Di Cristina; Oncologia Medica, Palermo, Sicily
  - La Maddalena Casa Di Cura Di Alta Specialita; Oncologia Chirurgica, Palermo, Sicily
  - Az. Osp. ; Divisione Di Oncologia, Ragusa, Sicily
  - Ospedale S. Croce Di Fano; Servizio Oncologia, Fano, The Marches
  - Ospedale Santa Chiara; Oncologia Medica, Trento, Trentino-Alto Adige
  - USL 8 Ospedale San Donato; Oncology Endocrinology, Arezzo, Tuscany
  - Ospedale Santa Maria Annunziata; Oncologia, Bagno a Ripoli, Tuscany
  - Azienda Ospedaliero-Universitaria Careggi;S.C. Oncologia Medica 1, Florence, Tuscany
  - Ospedale Campo Di Marte; Dipartimento Oncologico, Lucca, Tuscany
  - Azienda Usl 7; Dept. Oncologico, Poggibonsi, Tuscany
  - Arcispedale S.Anna; Oncologia Medica, Cona (Ferrara), Veneto
  - Polo Ospedaliero Santorso, Santorso, Veneto
  - Ospedale Civile S. Bortolo; Divisione Di Oncologia, Vicenza, Veneto
- Poland (2):
  - Regionalne Centrum Onkologi; Oddzial Chorob Wewnetrznych I Onkologii, Bydgoszcz
  - Oddzial Chemioterapii Szpitala Klinicznego Nr 1 w Poznaniu, Poznan
- Spain (9):
  - Hospital General de Mataro; Servicio de Oncologia, Mataró, Barcelona
  - Corporacio Sanitaria Parc Tauli; Servicio de Oncologia, Sabadell, Barcelona
  - Hospital de Navarra; Servicio de Oncologia, Navarra, Navarre
  - Hospital Universitario de Canarias;servicio de Oncologia, San Cristóbal de La Laguna, Tenerife
  - Complejo Hospitalario de Jaen-Hospital Universitario Medico Quirurgico; Servicio de Oncologia, Jaén
  - Hospital Regional Universitario Carlos Haya, Málaga
  - Hospital Universitario Virgen del Rocio; Servicio de Oncologia, Seville
  - Complejo Hospitalario de Toledo- H. Virgen de la Salud; Servicio de Oncologia, Toledo
  - Hospital Universitario Miguel Servet; Servicio Oncologia, Zaragoza
- Sweden (9):
  - Gävle sjukhus onkologkliniken, Gävle
  - Lanssjukhuset Ryhov; Onkologkliniken, Jönköping
  - Länssjukhuset Kalmar; Oncology, Kalmar
  - Centralsjukhuset Karlstad, Onkologkliniken, Karlstad
  - Uni Hospital Linkoeping; Dept. of Oncology, Linköping
  - Skånes University Hospital, Skånes Department of Onclology, Lund
  - Karolinska Hospital; Oncology - Radiumhemmet, Stockholm
  - Länssjukhuset Sundsvall, Onkologkliniken, Sundsvall
  - Norrlands Universitetssjukhus, Umeå, Cancercentrum; Dept of Oncology, Umeå
- United Kingdom (23):
  - Aberdeen Royal Infirmary; Medical Oncology Dept, Aberdeen
  - Belfast City Hospital; Dept of Oncology, Belfast
  - Velindre Cancer Centre; Oncology Dept, Cardiff
  - Broomfield Hospital; Oncology, Chelmsford
  - Ninewells Hospital; Dept of Radiotherapy & Oncology, Dundee
  - Royal Devon & Exeter Hospital; Oncology Centre, Exeter
  - Glasgow Western Infirmary; Dept of Radiotherapy, Glasgow
  - Huddersfield Royal Infirmary, Huddersfield
  - Queen Elizabeth Hospital, Kings Lynn
  - St Thomas Hospital; Medicine Div., London
  - St George'S Hospital; Oncology Research Office /Oncology Opd, London
  - Charing Cross Hospital; Medical Oncology., London
  - Christie Hospital; Breast Cancer Research Office, Manchester
  - James Cook Uni Hospital, Middlesbrough
  - Newcastle General Hospital, Newcastle upon Tyne
  - Royal Preston Hosptial, Preston
  - Oldchurch Hospital, Romford
  - Salisbury District General Hospital; Medical Oncology Dept, Salisbury
  - Royal Shrewsbury Hospitals Nhs Trust; Oncology, Shrewsbury
  - Southampton General Hospital; Medical Oncology, Southampton
  - Worthing Hospital; Sussex Oncology Centre, Worthing Breast Unit, Worthing
  - Yeovil District Hospital; Macmillan Cancer Unit, Yeovil
  - Airedale General Hospital; Oncology, York